CLINICAL TRIAL: NCT01610726
Title: Economic and Clinical Evaluation of Enhanced Recovery in Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010/2079
Record Dates: First submitted 2012-05-31; First posted 2012-06-04 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Colonic Diseases
Keywords: colon; rectum; recovery; surgery
MeSH Terms: conditions — Colonic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- enhanced recovery (Active Comparator)
  Interventions: Procedure: Enhanced versus conventional recovery in colorectal surgery
- conventional recovery (No Intervention)

INTERVENTIONS:
Procedure: Enhanced versus conventional recovery in colorectal surgery — Enhanced recovery (extended informations to the patients, change of anesthetic procedure, intravenous versus gas, and intensified mobilisation) versus conventional recovery
  Other Names: ERAS; Fast track surgery
  Arms: enhanced recovery

SUMMARY:
The purpose of this study is to evaluate the health cost and clinical outcome by introducing enhanced recovery (ERAS) compared to conventional recovery in colorectal surgery.

DETAILED DESCRIPTION:
Aim of the sudy:

1. Clinical evaluation: To investigate if patients treated with enhanced recovery have a shorter hospital stay and less morbidity than the patients treated conventionally. Other clinical questions witch might be answered in this study are clinical surgical stress response (insulin resistent), amount of analgetics used and time to normal activity.
2. Evaluation of quality of life: Instruments used in this sudy to evaluate quality of life are 15 D and qualitative interview.
3. Economic evaluation: Cost-utility analysis of the clinical studies
4. Compare patients who received a fast track program with dedicated fast track- and stoma nurse specialist and special focus on counselling and stoma education, compared with patients receiving existing current practice of stoma-education in a traditional care pathway, could reduce the length of hospital stay, readmission and stoma related complications
5. Further we will tray to generate additional insights into the impact of counselling when groups of patients are otherwise equal in terms of fast-track criteria. We are therefore continuing the enrolling of our colorectal patients in which both study arms contain the same ERAS items; the arms will only differ in terms of perioperative information and guidance as well as follow-up by dedicated nurses.

ELIGIBILITY:
Inclusion Criteria:

* Planed elective colorectal surgery, written consent and age above 18 years

Exclusion Criteria:

* Patients below 18 years, pregnancy, surgical emergency and no informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 484 (Actual)
Dates: Start 2012-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Length of stay | 30 days

SECONDARY OUTCOMES:
Morbidity | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Christian Erichsen, PhD, Study Chair — Helse Bergen, Haukeland University Hospital; Håvard Forsmo, MD, Study Chair — Helse Bergen, Haukeland University Hospital
Locations (1):
- Helse Bergen, Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Forsmo HM, Erichsen C, Rasdal A, Tvinnereim JM, Korner H, Pfeffer F. Randomized Controlled Trial of Extended Perioperative Counseling in Enhanced Recovery After Colorectal Surgery. Dis Colon Rectum. 2018 Jun;61(6):724-732. doi: 10.1097/DCR.0000000000001007. PMID 29664800